CLINICAL TRIAL: NCT05957653
Title: Lidocaine Combined With Sufentanil for Preventing Catheter-related Bladder Discomfort After Robot-assisted Radical Prostatectomy: a Randomized, Double-blind, Controlled Trial
Brief Title: Lidocaine Combined With Sufentanil for Preventing Catheter-related Bladder Discomfort
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, zhuhao, attending physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIT-2023-0092
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lidocaine; Sufentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine + sufentanil intervention group (Experimental)
  Interventions: Drug: lidocaine and sufentanil
- Saline control group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: lidocaine and sufentanil — A total of 20ml of 2% lidocaine and 1μg/ml sufentanil was injected into the bladder through the catheter.
  Arms: Lidocaine + sufentanil intervention group
Drug: Saline — A total of 20ml normal saline was injected into the bladder through the catheter.
  Arms: Saline control group

SUMMARY:
The goal of this clinical trial is to evaluate the incidence and severity of postoperative catheter-related bladder discomfort after robot-assisted radical prostatectomy.

The main question it aims to answer is to evaluate incidence of CRBD immediately after extubation in resuscitation.

A total of 20ml of 2% lidocaine and 1μg/ml sufentanil or 20ml normal saline was injected into the bladder of the participants through the catheter. After drug injection, the catheter was clamped for 20 minutes, and then 100ml normal saline was injected into the bladder through the catheter to flush out.

Then, the incidence of CRBD was compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-79 years, ASA class I-II
2. participants undergoing robot-assisted radical prostatectomy under general anesthesia
3. signed informed consent and volunteered to participate in the experiment

Exclusion Criteria:

1. urethral stricture, difficulty in inserting catheter or urethral bleeding during catheterization
2. a preexisting bladder disease such as an overactive bladder, bladder outflow obstruction, and neurogenic bladder
3. cognitive impairment or communication disorders
4. severe heart, lung, liver, kidney and immune system diseases
5. confirmed or suspected allergy to this trial drug

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
incidence of CRBD | immediately after extubation in resuscitation
  incidence of CRBD

IPD SHARING:
Plan to Share IPD: No